CLINICAL TRIAL: NCT06830551
Title: Personalized Approach in the Treatment of Patients Affected by Severe Dry Eye Associated With Therapy With EGFR Inhibitors (EGRFR-I) With Growth Factors in Cord Blood Serum (CBS) Eye Drops
Brief Title: The Effect of Cord Blood Serum Eyes Drops Administer in Patients With Severe Keratopathy Related to EGFR-I Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OFTAFONTANA_DED_EGFR-I; F35F22000080001 (Other Grant/Funding Number: Ministry of Health)
Record Dates: First submitted 2025-01-10; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-11

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eye drops derived from cordonal blood serum (Experimental): patients who are given eye drops
  Interventions: Drug: administration cord blood based eye drops, standardized to the deliver BDNF.

INTERVENTIONS:
Drug: administration cord blood based eye drops, standardized to the deliver BDNF. — administration cord blood based eye drops customized to deliver epitelio tropic factors, incluiding EGF in EGFR blocked cells

SUMMARY:
The study aim to evaluate the efficacy of cord blood eye drops in the healing of the damaged corneal epithelium.

DETAILED DESCRIPTION:
Patients undergoing treatment with EGFR inhibitor for lung cancer might develop corneal damage.

The study aims to evaluate the healing of corneal epithelium by administering cord blood eye drops for one month.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* oncology and advanced cancer patients who have EGFr mutation and who require treatment with antiEGFr drugs
* signing of informed consent

Exclusion Criteria:

* Patients who are unable to store/administer the CSCO independently, or with the help of care-givers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Corneal damage measured with National Eye Institute (NEI) score | one week before the start of treatment and thirty days after the end of treatment.
  Evaluation of the effect of cord blood eye drops administration on the variation of corneal damage in patients with severe keratopathy

SECONDARY OUTCOMES:
Change in discomfort | one week before the start of treatment and thirty days after the end of treatment.
  Symptomatology assessment with OSDI questionnaire. Quality of life analysis with Health-related SF-12 questionnaire, and SEI-QoL subjects' quality of life scale.
Change in quality of life | one week before the start of treatment and thirty days after the end of treatment.
  Change in QOL measured by SF-12 questionnaire
Change in quality of life | one week before the start of treatment and thirty days after the end of treatment.
  Change in QOL measured by SEI-QoL questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Fontana, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No